CLINICAL TRIAL: NCT04716231
Title: A Phase 2b/3, Multi-part, Randomized, Double-Blinded, Placebo-Controlled Study to Evaluate the Efficacy and Safety of Atacicept in Subjects With IgA Nephropathy (IgAN)
Brief Title: Atacicept in Subjects With IgA Nephropathy
Acronym: ORIGIN 3
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Vera Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: VT-001-0050
Record Dates: First submitted 2021-01-11; First posted 2021-01-20 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: IgA Nephropathy; Berger Disease
Keywords: Berger Disease; Berger's Disease; IGA Glomerulonephritis; IGA Nephropathy; Iga Nephropathy 1; Immunoglobulin A Nephropathy Nephritis; IGA Type Nephropathy, IGA
MeSH Terms: conditions — Glomerulonephritis, IGA | interventions — TACI receptor-IgG Fc fragment fusion protein

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Atacicept Dose 150mg (Experimental): Atacicept 150mg once weekly subcutaneous (SC) injections
  Interventions: Biological: Atacicept
- Placebo to match Atacicept (Part C/D) (Placebo Comparator): Placebo to match Atacicept once weekly subcutaneous (SC) injection
  Interventions: Other: Placebo to match Atacicept

INTERVENTIONS:
Biological: Atacicept — Once weekly subcutaneous (SC) injections by prefilled syringe
  Other Names: VT-001
  Arms: Atacicept Dose 150mg
Other: Placebo to match Atacicept — Once weekly subcutaneous (SC) injections by prefilled syringe
  Arms: Placebo to match Atacicept (Part C/D)

SUMMARY:
A Phase 3 Study with Atacicept in Subjects With IgA Nephropathy (ORIGIN 3)

DETAILED DESCRIPTION:
This is a multi-part study comprising of the original Phase 2b study and the addition of a separate pivotal Phase 3 study.

After the completion of the primary results for the Ph 2b dose ranging study, the pivotal study will evaluate the efficacy and safety of atacicept compared to placebo in reducing proteinuria in subjects with IgAN and persistent proteinuria despite being on a maximally tolerated dose (MTD) of a RASi. Safety, eGFR, serum immunoglobulins and Gd-IgA1 will also be clinically assessed. The clinical study is comprised of a 104wk double-blind treatment period, followed by a 52wk open-label treatment period and a 26wk safety follow-up period. The UPCR primary endpoint will be assessed after the first 200 patients are randomized.

ELIGIBILITY:
Key Inclusion Criteria:

* Must have the ability to understand and sign a written informed consent form
* Male or female of ≥18 years of age
* Total urine protein excretion ≥1.0 g per 24-hour or urine protein to creatinine ratio (UPCR) ≥1.0 mg/mg based on a 24-hour urine sample during the Screening Period
* Diagnosis of IgAN as demonstrated by renal biopsy conducted within 10 years
* eGFR ≥ 30 mL/min/1.73 m2, as per the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) equation.
* On a stable prescribed regimen of RAASi for at least 12 weeks that is at the maximum labeled or tolerated dose at Screening
* Systolic blood pressure ≤150 mmHg and diastolic blood pressure ≤90 mmHg

Key Exclusion Criteria:

* IgAN secondary to another condition (e.g., liver cirrhosis), or other causes of mesangial IgA deposition including IgA vasculitis (i.e., Henoch-Schonlein purpura), systemic lupus erythematosus (SLE), dermatitis herpetiformis, ankylosing spondylitis
* Total urine protein excretion ≥ 5g per 24-hour or urine protein to creatinine ratio (UPCR) ≥ 5 mg/mg based on a 24-hour urine sample during the Screening Period
* Evidence of rapidly progressive glomerulonephritis (loss of ≥ 50% of eGFR within 3 months of screening)
* Evidence of nephrotic syndrome within 6 months of screening (serum albumin <30g/L in association with UPCR >3.5 mg/mg
* Renal or other organ transplantation prior to, or expected during the study
* Concomitant chronic renal disease in addition to IgAN
* Uncontrolled diabetes, defined as hemoglobin-A1c (HbA1c) >7.5% at screening
* History of tuberculosis (TB), untreated latent TB infection (LTBI), or evidence of active TB determined by a positive Quantiferon test
* Participation in the Phase 2b (Parts A and B) study or any previous treatment with atacicept

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 376 (Estimated)
Dates: Start 2023-06-29 (Actual); Primary Completion 2025-05-15 (Actual); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in urine protein to creatinine ratio (UPCR) | 36 Weeks
  UPCR based on 24 hour urine collection

SECONDARY OUTCOMES:
Annualized rate of change in estimated glomerular filtration rate (eGFR) | 52 and 104 Weeks
  eGFR calculated by CKD-EPI formula

CONTACTS AND LOCATIONS:
Overall Officials: Zeeshan Khawaja, Study Director — Vice President, Clinical Development
Locations (1):
- ORIGIN 3 Global Site Contact Information, Brisbane, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Barratt J, Chen K, Lafayette R. A plain language summary: long-term safety and effectiveness of atacicept in individuals with IgA nephropathy. Curr Med Res Opin. 2026 Feb 1:1-15. doi: 10.1080/03007995.2026.2615321. Online ahead of print. PMID 41620980
- [Derived] Lafayette R, Barbour SJ, Brenner RM, Campbell KN, Doan T, Eren N, Floege J, Jha V, Kim BS, Liew A, Maes B, Pal A, Pecoits-Filho R, Phoon RKS, Rizk DV, Suzuki H, Tesar V, Trimarchi H, Wei X, Zhang H, Barratt J; ORIGIN Phase 3 Trial Investigators. A Phase 3 Trial of Atacicept in Patients with IgA Nephropathy. N Engl J Med. 2025 Nov 6. doi: 10.1056/NEJMoa2510198. Online ahead of print. PMID 41196369
- [Derived] Barratt J, Barbour SJ, Brenner RM, Cooper K, Wei X, Eren N, Floege J, Jha V, Kim SG, Maes B, Phoon RKS, Singh H, Tesar V, Lafayette R; ORIGIN Phase 2b Investigators. Long-Term Results from an Open-Label Extension Study of Atacicept for the Treatment of IgA Nephropathy. J Am Soc Nephrol. 2025 Apr 1;36(4):679-687. doi: 10.1681/ASN.0000000541. Epub 2024 Oct 26. PMID 39462308
- See also: Vera Therapeutics, Inc Company Website — http://www.veratx.com